CLINICAL TRIAL: NCT00735748
Title: Comparison of the Therapeutic Efficacy and Side Effects of Tramadol Per os (Tradonal Odis® Orodispersible Tablets) Versus an Optimised Dosis of Intravenous Tramadol for Postoperative Pain Relief in Ambulatory Surgery.
Brief Title: Comparison of Tramadol Orally Versus an Optimized Dose of Intravenous Tramadol for Postoperative Pain Relief in Ambulatory Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007/526
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Pain
Keywords: Patients who will undergo a general anesthesia for a procedure in short stay
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Tramadol per os (Tradonal Odis® orodispersible tablets)
  Interventions: Drug: Tramadol per os (Tradonal Odis® orodispersible tablets)
- 2 (Active Comparator): Tramadol IV (Tradonal® IV)
  Interventions: Drug: Tramadol IV (Tradonal® IV)

INTERVENTIONS:
Drug: Tramadol per os (Tradonal Odis® orodispersible tablets) — Administration of 1 unit dose of 50 mg tramadol perorally given in 3 unit dosages
  Arms: 1
Drug: Tramadol IV (Tradonal® IV) — Administration of tramadol IV given in 3 unit dosage of 35 mg
  Arms: 2

SUMMARY:
The purpose of this study is to compare the administration of 1 unit dose of 50 mg tramadol perorally given in 3 unit dosages versus tramadol IV given in 3 unit dosage of 35 mg during the first 6 hours postoperatively and to investigate the time course and accuracy of pain relief versus the onset and duration of side effects. The first unit dose will be administered at arrival at the PACU when a Visual Analogue Pain (VAS) score of more than 3 is reached. The second and third unit dose will be administered after 1 and 2 hours, respectively, when a VAS of more than 3 is observed.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II female or male patients undergoing wisdom teeth extraction
* Aged 18-70 years
* Scheduled for ambulatory surgery requiring postoperative pain medication

Exclusion Criteria:

* Weight less than 70% or more than 130% of ideal body weight
* Neurological disorder
* Recent use of psycho-active medication, including alcohol
* Patients suffering from chronic pain receiving pre-operative pain medication including NSAID's
* Use of chronic anti-emetic medication
* Use of chronic corticoid therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2008-03-01 (Actual); Primary Completion 2009-06-19 (Actual); Study Completion 2009-06-19 (Actual)

PRIMARY OUTCOMES:
Difference in pain score between groups | In the first hours after anaesthesia and surgery

SECONDARY OUTCOMES:
Difference in side-effects between the groups | In the first hours after anaesthesia and surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michel Struys, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be